CLINICAL TRIAL: NCT02572791
Title: Integrating Personal and Household Environmental Hygiene Measures to Prevent Methicillin-Resistant Staphylococcus Aureus Infection
Brief Title: Staph Household Intervention for Eradication (SHINE)
Acronym: SHINE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Stephanie A. Fritz, Professor of Pediatrics, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3177 60559
Record Dates: First submitted 2015-10-05; First posted 2015-10-09 (Estimated); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Skin and Subcutaneous Tissue Bacterial Infections; Staphylococcus Aureus; MRSA - Methicillin Resistant Staphylococcus Aureus Infection
MeSH Terms: conditions — Staphylococcal Infections | interventions — Chlorhexidine; chlorhexidine gluconate; Mupirocin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Periodic personal decolonization (Experimental): All household participants will perform chlorhexidine body washes twice weekly for 3 months and apply mupirocin ointment to the anterior nares twice daily for five consecutive days each month for 3 months.
  Interventions: Drug: Chlorhexidine; Drug: Mupirocin
- Household environmental hygiene (Experimental): In addition to their usual cleaning, households will be asked to perform targeted household hygiene focusing on sources known to harbor S. aureus and serve as reservoirs for transmission.
  Interventions: Behavioral: Household cleaning
- Integrated personal/household hygiene (Experimental): Participants in households randomized to this arm will perform the Periodic Personal Decolonization plus the Household Environmental Hygiene, described above in arms 1 and 2.
  Interventions: Drug: Chlorhexidine; Drug: Mupirocin; Behavioral: Household cleaning

INTERVENTIONS:
Drug: Chlorhexidine
  Other Names: Hibiclens
  Arms: Integrated personal/household hygiene; Periodic personal decolonization
Drug: Mupirocin
  Other Names: Bactroban
  Arms: Integrated personal/household hygiene; Periodic personal decolonization
Behavioral: Household cleaning
  Arms: Household environmental hygiene; Integrated personal/household hygiene

SUMMARY:
The investigators propose a pragmatic comparative effectiveness trial evaluating several decolonization strategies in patients with Staphylococcus aureus infection, their household contacts, and household environmental surfaces. The central hypothesis of this proposal is that an integrated approach of periodic personal and household environmental hygiene will reduce S. aureus transmission in households and subsequently decrease the incidence of skin and soft tissue infections (SSTI).

DETAILED DESCRIPTION:
Patients with active or recent S. aureus SSTI will be recruited from St. Louis Children's Hospital and community pediatric practices affiliated with the investigators practice-based research network. All participants (index patients and their household contacts) will perform a baseline S. aureus decolonization protocol for 5 days consisting of enhanced hygiene measures, application of mupirocin antibiotic ointment to the anterior nares twice daily, and daily body washes with chlorhexidine antiseptic. Following the 5-day baseline decolonization regimen, households will be randomized to one of three intervention groups: 1) Periodic personal decolonization performed by all household members, to include chlorhexidine body washes twice weekly for 3 months and application of intranasal mupirocin for 5 consecutive days each month for 3 months; 2) Household environmental hygiene, including targeted cleaning of household surfaces and laundering of bed linens, weekly for 3 months; and 3) Integrated periodic personal decolonization and household environmental hygiene for 3 months. Households will be followed prospectively (1, 3, 6, and 9 months following randomization) to measure the prevalence of S. aureus colonization in the participants, household environmental surfaces, and pet dogs and cats and to document the incidence of recurrent SSTI. Molecular strain typing will be performed on all recovered S. aureus isolates to illuminate transmission dynamics and the effects of the decolonization measures on genetic epidemiology. Lastly, the investigators will assess resistance to the prescribed topical antimicrobials at baseline and longitudinal samplings.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age and younger
* Confirmed (i.e., culture-positive) active or recent (within the past 2 months) S. aureus cutaneous infections
* Reside within 75 miles of St. Louis Children's Hospital
* Provide written, informed consent, or consent is provided by a parent or legal guardian

Exclusion Criteria:

* Patients with nosocomial infections (i.e., >48 hours after hospitalization)
* Patients with traditional risk factors for HA-MRSA (e.g., immunodeficiency, indwelling catheter or percutaneous medical device, undergoing dialysis, presenting with a surgical site infection, or residing in a long-term care facility within the past year).
* Patients who are unable to give consent or for whom consent is not obtained
* Patients refusing home environmental cultures by the study team
* Patients without a permanent home (e.g., living in a shelter or group home)

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 835 (Actual)
Dates: Start 2015-10; Primary Completion 2024-11 (Actual); Study Completion 2024-12 (Actual)

PRIMARY OUTCOMES:
Incidence of SSTI | 3 months after randomization
  We will compare the incidence of SSTI at the household level (i.e., occurring in any household member) 3 months after randomization between the Integrated Decolonization Group and the combined Personal Periodic Decolonization and Environmental Decontamination Groups.

SECONDARY OUTCOMES:
Prevalence of S. aureus colonization in index patients, household contacts, pet dogs and cats, and household surfaces | 9 months (collected at baseline, 1 month, 3 months, 6 months, and 9 months).
  Describe baseline and longitudinal prevalence of MRSA colonization in index patients, household contacts, pet dogs and cats, and household surfaces and compare between the 3 intervention groups.
Confirmed S. aureus Infection | 9 months
  We will compare the development of a confirmed S. aureus infection between participants in the 3 groups over 9 months at the household and individual level.
Number of patients with adverse events due to study intervention | 3 months
  We will describe the number of participants with adverse events due to study intervention (e.g., rhinorrhea, rash, dry skin) and compare between the three groups.
Mupirocin resistance | 9 months
  Measure the prevalence of mupirocin resistance in S. aureus strains recovered at serial samplings over the study period of 9 months.
Number of participants adhering to study intervention procedures | 3 months
  We will describe the number of participants completing chlorhexidine baths, mupirocin applications, and household hygiene measures.
Incidence of SSTI | 1 month, 6 months, and 9 months after randomization
  We will compare the incidence of SSTI at the household level (i.e., occurring in any household member) 1 month, 6 months, and 9 months after randomization between the Integrated Decolonization Group and the combined Personal Periodic Decolonization and Environmental Decontamination Groups.
  In addition to to the household level, we will also assess SSTI outcomes at the individual household member level, the index patient level, and the household contact level.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie A Fritz, MD, MSCI, Principal Investigator — Washington University School of Medicine
Locations (2):
- United States (2):
  - St. Louis Children's Hospital, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri